CLINICAL TRIAL: NCT03320681
Title: Effect Mechanism of a Non-invasive Stimulation Device for Rapid Alleviation of Parkinson's Disease Symptoms
Brief Title: Effect Mechanism Investigation of a Non-invasive Stimulation Device for Rapid Alleviation of Parkinson's Disease Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inventram (Industry)
Collaborators: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Par-02
Record Dates: First submitted 2017-08-16; First posted 2017-10-25 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
Keywords: Neurostimulator
MeSH Terms: conditions — Parkinson Disease | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation (Active Comparator): Acupuncture needles will be inserted into the auricular zones and electrical stimulation will be given for 20 minutes.
  Interventions: Device: Electrical Stimulation
- Dry Needling (Other): Acupuncture needles will be inserted into the auricular zones for 20 minutes. However, no electrical stimulation will be given
  Interventions: Other: Dry Needling Stimulation

INTERVENTIONS:
Device: Electrical Stimulation — Percutaneous electrical nerve stimulation
  Arms: Active Stimulation
Other: Dry Needling Stimulation — Percutaneous nerve stimulation
  Arms: Dry Needling

SUMMARY:
Effect Mechanism Investigation of a Wearable Electrostimulator for Rapid Alleviation of Parkinson's Disease Symptoms

DETAILED DESCRIPTION:
Activation levels of interested regions of the brain will be measured through fMRI technique prior and after the dry needling and active stimulation applications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* H&Y Stage >= 2
* Existing bradykinesia symptoms
* Existence of one of the symptoms below
* Resting Tremor
* Rigidity
* Walking disorder

Exclusion Criteria:

* Cardiac Pacemaker
* Psychiatric diagnosis
* Irregular heart/respiration rate
* Pregnancy
* Alcohol consumption
* Cardiovascular disease history
* Wearing an electro-active prosthesis
* Brain surgery history
* Ongoing TENS/PENS therapy-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
fMRI - Activation level comparison of the motor and supplementary cortex | Baseline and PostStim (right after the stimulation is terminated)
fMRI - Activation level comparison of the subthalamic nucleus (STN) and basal ganglia including pedunculopontine nucleus (PPN) | Baseline and PostStim (right after the stimulation is terminated)
fMRI - STN, PPN and cortical connectivity alterations | Baseline and PostStim (right after the stimulation is terminated)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf O Cakmak, Phd, MD, Principal Investigator — Otago University; Burak Ozsoy, PhD, Study Director — Inventram
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No